CLINICAL TRIAL: NCT04549103
Title: Effect of Community-based Baduanjin (八段锦) on Functional Performance in Pre-Frail/Frail Older Adults: A Randomised Controlled Trial
Brief Title: Effect of Baduanjin on Functional Performance in Pre-Frail/Frail Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geriatric Education and Research Institute (Other Government)
Collaborators: Tsao Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCMG BDJ RCT
Record Dates: First submitted 2020-08-24; First posted 2020-09-16 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Frailty; Frail Elderly Syndrome
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention group will receive the 16-week Baduanjin exercise intervention.
  Interventions: Other: Baduanjin exercise program
- Control Group (No Intervention): Control group will not receive the exercise intervention, but they will attend four education classes about managing their health status.

INTERVENTIONS:
Other: Baduanjin exercise program — Baduanjin (BDJ), also known as Eight-Section Brocades, is one of the forms of traditional Chinese Qigong exercises, characterized by symmetrical physical posture, movements, mindfulness, and breathing. Its primary focus is on the release of 'Qi' or internal body energy with the intent of improving health outcomes. BDJ encompasses eight simple movements involving combinations of postures, meditation, slow relaxing movements, and breathing exercises. It is a low intensity exercise, which have been found to improve range of motion, strength and general health. The simplicity and low intensity level is ideal for older adults to practice at home using instructional videos.
  Arms: Intervention Group

SUMMARY:
The aim for this study is to investigate the effectiveness of a 16-week realistic community-delivered Baduanjin training program compared to a waitlist control intervention, in improving functional outcomes among pre-frail and frail older adults in Singapore. It is hypothesized that participants that receive 16-week of BDJ training will have significant improvement in physical function (including balance, muscle strength, and endurance); alleviate exhaustion; reduce risk of falling and fear of falling; potentially reverse frailty; reduce depression; and improve quality of life, potentially with greater improvements in area(s) for individuals with lower baseline measures. Whereas, participants in the waitlist control group, will have insignificant changes to their baseline measures.

ELIGIBILITY:
Inclusion Criteria:

* Pre-frail and frail adults aged 55 years and above
* Able to ambulate (move about) without personal assistance and has no other physical limitations affecting participation and adherence
* Able to understand basic instructions
* Generally sedentary lifestyle

Exclusion Criteria:

* Participating in other intervention studies
* Perform regular moderate to vigorous intensity exercise
* Perform regular Taichi or Qigong exercise
* Have severe audio-visual impairment
* Diagnosed with cognitive impairment (e.g. dementia, Alzheimer's Disease) and/or history of neurological disorder (e.g. cerebral palsy, Parkinson's Disease)
* Diagnosed with postural hypotension (have a drop of 20mmHg systolic blood pressure, or a drop of 10mmHg diastolic blood pressure within two to five minutes of standing up, or if standing causes signs and symptoms)
* Unable to participate for the full duration of the study
* Unable to come to the training site by himself/herself or by the help of caregivers
* Not suitable to participate in exercise as deemed by a medical doctor

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Change in Knee Extension Strength | Baseline, and after 16-weeks of intervention
  Knee extension strength is measured using a digital dynamometer gauge. Prior to performing the test, leg dominant is determined by asking participants which is their dominant leg or which leg they would predominantly use when performing a task. For the assessment, participants will be asked to extend their leg against the spring gauge while seated with the hip and knee joint angles positioned at 90°. Maximal force is recorded in kilograms.
Change in Maastricht Vital Exhaustion Score (MQ) | Baseline, and after 16-weeks of intervention
  Maastricht vital exhaustion score (MQ) is a short questionnaires that requires between 5 to 10 minutes for completion. MQ is a validated tool to assess feelings of "vital exhaustion", which has three defining characteristics: (1) feeling of excessive fatigue and lack of energy, (2) increased irritability, and (3) feelings of demoralization.
Change in Falls Efficacy Scale-International (FES-I) | Baseline, and after 16-weeks of intervention
  The Falls Efficacy Scale-International (FES-I) is a short, easy to administer tool that measures the fear of falling in older population during social and physical activities inside and outside the home. The level of concern is measured on a four point Likert scale (1=not at all concerned to 4=very concerned). The 16-item FES-I is a well validated and feasible measure to assess fear of falling in older persons, and predicts future risks of falls.

SECONDARY OUTCOMES:
Change in Physiological Profile Assessment. (PPA - Short Form) | Baseline, and after 16-weeks of intervention
  Physiological Profile Assessment (PPA) is a valid and reliable measure of balance function and fall risk, is feasible for older adults to undertake, and can quantify changes in specific physical components contributing to falls in response to BDJ training. PPA comprises a series of five sensorimotor assessments: edge contrast sensitivity, lower limb proprioception, knee extension strength, hand reaction time, and postural sway. These five components will be weighted to compute a composite PPA fall risk score: high composite PPA scores indicate high risk of falling.
Change in Hand Grip Strength | Baseline, and after 16-weeks of intervention
  Hand-grip dynamometer was found to be a valid tool in clinical and research practice, and is an easy, quick, and inexpensive way of assessing HGS in older adults. Prior to performing the hand-grip strength test, hand dominance is determined by asking participants which hand they use for writing or which hand they would predominantly use when performing a task. HGS is measured in kilograms by taking the average of the two dominant handgrip attempts using a Jamar Plus + Digital Hand Dynamometer.
Change in 6-meter Fast Gait Speed Test | Baseline, and after 16-weeks of intervention
  The purpose of the gait speed test is to measure the participant's fastest speed while walking and mobility. Fast gait speed is determined across a distance of 6 meter, which is marked on the floor with tape. Subjects are allowed to use their usual walking aid. Two trails will be administered, time (in seconds) will be recorded for each trial. The average speed of two trails will be recorded as the fast gait speed.
Change in Time Up and Go test (TUG) | Baseline, and after 16-weeks of intervention
  Time Up and Go test (TUG) is a reliable and valid test for quantifying functional mobility for frail elder person. The participant is observed and timed while he rises from an arm chair, walks 3 meters, turns, walks back, and sits down again. As the test is quick, and requires no special equipment or training, it is widely used in studies as a physical assessment.
Change in 30 seconds Sit-to-stand (STS) | Baseline, and after 16-weeks of intervention
  Sit-to-stand (STS) test is a commonly used functional performance measure in clinical research and practice. STS performance is influenced by multiple physiological and psychological processes and represents a particular transfer skill, rather than a proxy measure of lower limb strength. In 30 seconds STS, participants will be asked to rise from the chair as fast as possible with their arms fold across their chest and the number of times they are able to perform sit-to-stand successfully within 30 seconds will be recorded. The performance of this test is suggested to be influenced by factors associated with balance, muscle strength, lower extremity endurance, and mobility as well.
Change in Frailty Score | Baseline, and after 16-weeks of intervention
  Frailty score of the participants will be assessed based on the five criteria by Fried in the Cardiovascular Health Study (CHS). The five criteria (modified for this pilot study) include: unintentional weight loss >10 lbs (4.5kg) and/or BMI of <18.5 in the last 6 months measured by self-report, weakness measured by knee extension strength, slowness measured by 6-m gait speed, exhaustion measured by questionnaire (SF-12), and physical inactivity measured by LASA Physical Activity Questionnaire. One-point is assign for the presence of each component, and based on the individual's total score, participants are categorized as frail (3-5 points), pre-frail (1-2 points), and robust (0 point). Reduction in frailty during the study is defined as a transition to a lower frailty category from baseline over 3 months.
Change in EuroQol-Five Dimensions (EQ-5D) | Baseline, and after 16-weeks of intervention
  EQ-5D is one of the most commonly used generic health quality of life (QoL) status measurement, and its good validity and reliability have been reported in various health conditions. In this study, EQ-5D will be used as a standardized instrument for measuring generic health-related QoL.
Change in Geriatric Depression Scale (GDS) | Baseline, and after 16-weeks of intervention
  GDS is a 30-item self-report assessment used to identify depression in the elderly. One point is assigned to each answer and the cumulative score is rated on a scoring grid. The grid sets a range of 0-9 as "normal", 10-19 as "mildly depressed", and 20-30 as "severely depressed".

CONTACTS AND LOCATIONS:
Locations (1):
- Yong-en Care Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu X, Seah JWT, Pang BWJ, Tsao MA, Gu F, Ng WC, Tay JYR, Ng TP, Wee SL. A single-arm feasibility study of community-delivered Baduanjin (Qigong practice of the eight Brocades) training for frail older adults. Pilot Feasibility Stud. 2020 Jul 21;6:105. doi: 10.1186/s40814-020-00649-3. eCollection 2020. PMID 32699644
- [Derived] Tou NX, Goh SF, Harding S, Tsao MA, Ng TP, Wee SL. Effectiveness of community-based Baduanjin exercise intervention for older adults with varying frailty status: a randomized controlled trial. Eur Rev Aging Phys Act. 2024 Oct 10;21(1):28. doi: 10.1186/s11556-024-00363-6. PMID 39390362